CLINICAL TRIAL: NCT07285902
Title: A Multicenter, Randomized, Open-label, Parallel-controlled Phase III Study Comparing the Efficacy and Safety of HRS9531 Injection Versus Semaglutide Injection in Subjects With Obesity
Brief Title: A Study Comparing the Efficacy and Safety of HRS9531 Injection With Semaglutide Injection in Subjects With Obesity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-308
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: HRS9531 injection (Experimental)
  Interventions: Drug: HRS9531 injection
- Treatment group B: Semaglutide Injection (Active Comparator)
  Interventions: Drug: Semaglutide Injection

INTERVENTIONS:
Drug: HRS9531 injection — HRS9531 injection
  Arms: Treatment group A: HRS9531 injection
Drug: Semaglutide Injection — Semaglutide Injection
  Arms: Treatment group B: Semaglutide Injection

SUMMARY:
This study is a multicenter, randomized, open-label, parallel-controlled, phase III study to compare the efficacy, safety, and tolerability of HRS9531 versus semaglutide once weekly (QW) in adult subjects with obesity

ELIGIBILITY:
Inclusion Criteria:

1. With my consent and has signed the informed consent form, I am willing and able to follow the requirements of the trial protocol to complete this study;
2. Age ≥ 18 years old on the day of signing the informed consent, regardless of gender;
3. obesity
4. Self-reported diet and exercise control for 3 months or more before screening, and weight change of ≤ 5 kg in the past 3 months.
5. Male and female subjects of childbearing potential (including partners) who have no fertility plan and agree to take highly effective contraceptive measures within 2 months after signing the informed consent form to the last dose, and female or male subjects of childbearing potential have no plans to donate eggs/sperm; Female subjects of childbearing potential have a negative pregnancy test within 3 days prior to randomization and are not lactating.

Exclusion Criteria:

1. Those with abnormal relevant examinations at screening;
2. ECG results are abnormal and may affect the safety of the subject
3. Poor blood pressure control
4. The PHQ-9 score ≥ 15 points
5. Presence or history of endocrine disorders that may significantly affect body weight
6. History of diabetes mellitus
7. Those who have had any previous disease or history that affects gastric emptying, or who have undergone gastrointestinal surgery
8. Previous or known history of acute or chronic pancreatitis, pancreatic injury; Patients with a history of acute cholecystitis or symptomatic/treatment-inducing gallbladder disease
9. Previous or known history or family history of medullary thyroid cancer (MTC) or multiple endocrine neoplasia type 2 (MEN2).
10. Severe infection, severe trauma, or large and medium-sized surgery within 1 month prior to screening
11. History of severe cardiovascular and cerebrovascular diseases within the previous 6 months
12. Malignancy of any organ system within 5 years
13. Presence or suspicion of depression, bipolar disorder, suicidal tendencies, People with schizophrenia or other more serious mental illness
14. Known or suspected history of alcohol and/or drug abuse or drug abuse
15. Presence of a history of acute or chronic hepatitis or other serious liver disease other than non-alcoholic fatty liver disease
16. Presence of any hematologic disorder that may interfere with HbA1c detection
17. Presence of autoimmune disease with planned use of systemic glucocorticoids or immunosuppressive therapy during the study
18. Use of medications or treatments that may result in significant weight gain or loss within the previous 3 months
19. Received, or planned to undergo bariatric surgery or endoscopic and/or medical device-based bariatric therapy during the study, etc
20. Those who have a known or suspected allergy to the same or related products of the investigational drug and their excipients
21. Previous discontinuation of this class for safety/tolerability reasons
22. Participation in a clinical trial of any drug or medical device within 3 months prior to screening
23. Those who have donated or lost ≥ 400 mL of blood within the previous 3 months, or have received blood transfusions
24. Surgery is planned for the duration of the trial
25. Subjects who are mentally incapacitated or have language impairment who are unable to fully understand or participate in the trial process
26. Investigators and relevant staff of the research center or other persons directly involved in the implementation of the program, and their immediate family members; Employees of Hengrui Company; In the judgment of the investigator, there is any condition that affects the safety of the subject or any other interference with the evaluation of the test results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in body weight after 52 weeks of treatment | 52 weeks

SECONDARY OUTCOMES:
Proportion of subjects with target reduction from baseline in body weight after 52 weeks of treatment | 52 weeks
Change from baseline in waist circumference,after 52 weeks of treatment | 52 weeks
Change from baseline in body weight after 52 weeks of treatment | 52 weeks
Change from baseline in body mass index (BMI) after 52 weeks of treatmentChange from baseline in blood pressure,after 52 weeks of treatment | 52 weeks
Change from baseline in fasting plasma glucose (FPG)after 52 weeks of treatment | 52 weeks
Change from baseline in glycosylated haemoglobin (HbA1c) after 52 weeks of treatment | 52 weeks
Change from baseline in liver enzymes after 52 weeks of treatment | 52 weeks
Change from baseline in fasting serum insulin after 52 weeks of treatment | 52 weeks
Change from baseline in lipid parameters after 52 weeks of treatment | 52 weeks
Number of AEs during the trial. | 52 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chiness PLA General Hospital, Beijing, Beijing Municipality
  - Jiangsu Province Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided